CLINICAL TRIAL: NCT07286032
Title: A Randomized, Multi-Center, Double-Blind, Phase III Study Evaluating the Efficacy and Safety of Hetrombopag Olamine Tablets Vs Placebo in Patients With Chemotherapy-Induced Thrombocytopenia
Brief Title: A Study to Evaluate the Efficacy and Safety of Hetrombopag Olamine Tablets Vs Placebo in Patients With Chemotherapy-Induced Thrombocytopenia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8735-303
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Patients With Chemotherapy-Induced Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Hetrombopag Olamine (Experimental)
  Interventions: Drug: Hetrombopag Olamine
- Part B：Hetrombopag Olamine vs Hetrombopag Olamine Placebo (Experimental)
  Interventions: Drug: Hetrombopag Olamine ；Hetrombopag Olamine Placebo

INTERVENTIONS:
Drug: Hetrombopag Olamine — For Part A, all participants would receive hetrombopag treatment.
  Arms: Part A: Hetrombopag Olamine
Drug: Hetrombopag Olamine ；Hetrombopag Olamine Placebo — For Part B，participants would be randomized to receive hetrombopag treatment or matching placebo, respectively。
  Arms: Part B：Hetrombopag Olamine vs Hetrombopag Olamine Placebo

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of of Hetrombopag Olamine Tablets Vs Placebo in Patients with Chemotherapy-Induced Thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female gender, age ≥18 years at screening.
2. Histologically or cytologically confirmed solid tumor (e.g., non-small-cell lung carcinoma [NSCLC], breast, ovarian, bladder, pancreatic, gastrointestinal, or colon/colorectal cancer).
3. Receiving platinum- and/or gemcitabine-containing chemotherapy regimens on 21-day treatment cycles.
4. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
5. Life expectancy ≥6 months.
6. Signed ICF for voluntary participation in the study and good compliance.

Exclusion Criteria:

1. Hematopoietic diseases other than CIT (e.g., primary immune thrombocytopenia).
2. Hematologic malignancies.
3. Thrombocytopenia caused by reasons other than chemotherapy, including but not limited to chronic liver disease, hypersplenism, infection, and hemorrhage, within 6 months prior to Study Day 1.
4. Untreated brain metastases; or with leptomeningeal metastasis.
5. Conditions that require emergent treatment (e.g., superior vena cava syndrome, spinal cord compression).
6. Severe cardiovascular disorders or interventions within 6 months
7. Have arterial/venous thrombosis within 6 months
8. Known bleeding disorders, platelet dysfunction
9. Severe haemorrhage during screening
10. Acute or uncontrolled hepatitis B&C infection
11. Human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Part A: Cmax of hetrombopag in non-Asian participants with CIT, around 6 months. | around 6 months.
Part A: AUC0-tauof hetrombopag in non-Asian participants with CIT, around 6 months | around 6 months
Part A: Cmin of hetrombopag in non-Asian participants with CIT, around 6 months | around 6 months
Part B:A platelet count of ≥100×109/L within 14 days after initiating the investigational product treatment, around 3 years | around 3 years
Part B:No use of any rescue therapy for thrombocytopenia during the treatment period from the initiation of investigational product treatment until Cycle 2 Day 21, around 3 years. | around 3 years.
Part B:Complete two consecutive on-study chemotherapy cycles (Cycle 1 and Cycle 2) without thrombocytopenia-induced modification of any myelosuppressive agent, around 3 years; | around 3 years;

SECONDARY OUTCOMES:
Proportion of participants achieving platelet count ≥100×109/L without the use of rescue therapy within 14 days after initiating the investigational product treatment,around 3 years; | around 3 years;
platelet count nadir from Cycle 1 Day 1 until Cycle 2 Day 21, around 3 years; | around 3 years;
Proportion of participants free from serious bleeding events, during the treatment period from the initiation of IP treatment until C2D21, around 3 years; | around 3 years;
Proportion of participants with neutropenia during the treatment period from the initiation of IP treatment until Cycle 2 Day 21, around 3 years. | around 3 years.
Number of Adverse Events/Serious Adverse Events, safety lab parameters, vital signs, etc within study period, around 3 years. | around 3 years.

IPD SHARING:
Plan to Share IPD: Undecided